CLINICAL TRIAL: NCT04468230
Title: Phase 2 Study of Nicotine for the Treatment of Pain Associated With Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Study of Nicotine for Pain Associated With Chemotherapy-Induced Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual Rate
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-16-12518
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Neuropathy; Peripheral Neuropathy; Neuropathic Pain; Chemotherapy-induced Peripheral Neuropathy
Keywords: Nicotine; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine Transdermal Patch Administration (Experimental): Each patient will complete two 14-day treatment conditions, for 7 mg nicotine transdermal patch administration with a washout period in between (≥ 14 days and up to 21 days), then 14 mg nicotine transdermal patch administration (14 days).
  Interventions: Drug: Nicotine Transdermal Patch

INTERVENTIONS:
Drug: Nicotine Transdermal Patch — Nicotine Treatment Condition

SUMMARY:
Assess the efficacy of short-term nicotine transdermal patch administration for the treatment of chemotherapy-induced peripheral neuropathy (CIPN) in cancer stable patients or patients in remission.

DETAILED DESCRIPTION:
This phase 2 study will test the efficacy of short-term transdermal nicotine transdermal patch administration in patients who have been diagnosed with CIPN. The study will follow an open-label, crossover within-subjects clinical trial design with nicotine transdermal patch.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed peripheral sensory neuropathy defined as:
* Greater than Grade 1 peripheral sensory neuropathy using the CTCAE v5.0 grading scale

  * Grade 1 Asymptomatic
  * Grade 2 Moderate symptoms; limiting instrumental activities of daily living (ADL)
  * Grade 3 Severe symptoms; limiting self-care ADL
  * Grade 4 Life-threatening consequences; urgent intervention indicated
* Have a baseline chemotherapy-induced peripheral neuropathy (CIPN) patient reported outcome (PRO) total sensory score ≥ 24.3 on a 19 to 76 scale using the European Organization for Research and Treatment of Cancer Quality of Life-CIPN20 Questionnaire (EORTC QLQ-CIPN-20)
* Have a CIPN-related neuropathic pain score ≥ 4 on a 0 to 10 scale using the Brief Pain Inventory-Short Form (BPI-SF) item 5
* Will not have used any nicotine or tobacco products (eg, cigarettes, electronic cigarettes, smokeless tobacco, or other nicotine replacement therapies) within 14 days prior to study treatment start date
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Not currently receiving any chemotherapy
* Have previously received platinum- and/or taxane-based chemotherapy treatments and have persistent pain at least 3 months after completion of treatments.
* Willing and able to comply with study procedures and visit schedule.
* Willing to abstain from all tobacco/nicotine product use during study treatment and 30-day follow-up period.
* Ability to self-apply or have the patch applied at home daily.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of pre-existing peripheral sensory neuropathies related to the following:

  * Autoimmune disease
  * B12/folate deficiency
  * Diabetes Mellitus
  * Human immunodeficiency virus (HIV)
  * Hyper/hypothyroidism
  * Monoclonal gammopathy of undetermined significance or multiple myeloma
* History of receiving other types of neurotoxic chemotherapy drugs (eg, vinca alkaloids, bortezomib, thalidomide)
* Current or prior pheochromocytoma
* History of or active or clinically significant cardiac disease including any of the following:

  * Unstable angina (eg, anginal symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
  * Myocardial infarction diagnosed within 6 months prior to initiating study treatment
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers
* New York Heart Association (NYHA) class III or IV congestive heart failure
* Poorly controlled high or low blood pressure defined as:

  * Systolic blood pressure (SBP) ≥ 140; Diastolic blood pressure (DBP) ≥ 90
  * SBP ≤ 90; DBP ≤ 60
* Regular use of the following medications:

  * Varenicline
  * Bupropion (ie, bupropion hydrochloride sustained release)
* Women will be excluded if they are breastfeeding or are pregnant (by urinalysis) within 14 days prior to the start of nicotine transdermal patch administration.
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, MD, Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Virginia Commonwealth University, Richmond, Virginia
  - VCU Community Memorial Healthcenter, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotine Transdermal Patch Administration
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Confidentiality is an issue.
Arm/Group | Nicotine Transdermal Patch Administration
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Short-term Nicotine Transdermal Patch Administration in the Treatment of Cancer Induced Peripheral Neuropathy (CIPN)
Description: To assess the efficacy, of the nicotine transdermal patch administration in the treatment of CIPN in patients whose cancer is stable or in remission as defined by a ≥ 2.7 point decrease in the total sensory score of the European Organization for Research and Treatment of Cancer Quality of Life-cancer induced peripheral neuropathy (CIPN20) Questionnaire (EORTC QLQ-CIPN-20) (eg, an improvement in the patients quality of life by one grade). The QLQ-CIPN20 numerical score has a range of 19-76, in which lower scores indicate less symptoms and a better quality of life.
Time Frame: 79 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Transdermal Patch Administration
Number analyzed (Participants) | 3
score on a scale
  7mg patch | -7.7 (10.5)
  14 mg patch | -2.0 (5.0)

2. Secondary Outcome: Efficacy of Pain-related Changes and Degree of Functional Interference in the Treatment of CIPN
Description: To assess the efficacy of short-term nicotine transdermal patch administration in the treatment of CIPN in patients whose cancer is stable or in remission by assessing changes in the degree of pain-related functional interference measured by the Brief Pain Inventory - Short Form (BPI-SF) interference score. The BPI-SF contains 4 items assessing average, worst, least, and immediate pain severity in the last 24 hours. Pain severity items are scored using an 11-point numeric rating scale (0, no pain; 10, pain as bad as you can imagine). Seven BPI-SF items will be used to quantify the degree to which pain interferes with daily activities or function (0, does not interfere; 10, completely interferes). The 7 items are summed to obtain a total interference score.
Time Frame: 79 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Transdermal Patch Administration
Number analyzed (Participants) | 3
score on a scale
  7 mg patch | -1.3 (2.1)
  14 mg patch | -2.0 (1.7)

3. Secondary Outcome: Number of Participants at Risk and Affected by Adverse Events (AEs) Related to the Transdermal Nicotine Patch.
Description: To assess the AEs profile of nicotine transdermal patch administration for the treatment of CIPN in patients whose cancer is stable or in remission. The Adverse events (AEs) are reported using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version (CTCAE v 5.0)
Time Frame: 79 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Transdermal Patch Administration
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: All adverse events (AE's) regardless of grade or attribution will be recorded from the beginning of study treatment (Cycle 1, Day 1 of nicotine transdermal patch administration) through the 30-day follow-up period.
Arm/Group | Nicotine Transdermal Patch Administration
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Transdermal Patch Administration (N=4)
Sinus Tachycardia (Cardiac disorders) | 1 (2)
Eye disorders- other (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5)
Headache (Nervous system disorders) | 3 (6)
Nervous System Disorders, Other (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
The Coronavirus-19 (COVID-19) pandemic caused reduced accrual rates. The protocol was terminated early due to slow accrual rates by the Protocol Review & Monitoring Committee (PRMC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04468230/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04468230/ICF_001.pdf